CLINICAL TRIAL: NCT05797194
Title: The Potential Value of Systemic Inflammation Response Index on Postoperative Delirium in Older Patients
Brief Title: The Association Between SIRI and POD in Older Patients
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: POD-SIRI
Record Dates: First submitted 2023-03-05; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Delirium; Elderly; Surgery
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POD group: Patients were considered to surfer from postoperative delirium by a positive Confusion Assessment Method (CAM) questionnaire after surgery.
- No-POD group: Patients did not surfer from postoperative delirium by a positive CAM questionnaire after surgery.

SUMMARY:
Postoperative delirium (POD) remains one of most common complication in elderly patients receiving surgery, which is characterized by acute and fluctuating change in the level of cognition and consciousness. Previous studies have shown that surgery and anesthesia-induced acute peripheral inflammation and neuroinflammation may lead to delirium after surgery. Systemic Inflammation Response Index (SIRI) is a more easily accessible and comprehensive inflammation marker derived from monocyte, neutrophil, and lymphocyte count, which has been investigated to assess the prognosis of cancer and infectious diseases. However, the relationship between SIRI and POD has yet to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Hospital stay of at least 3 days
* More than or equal to 65 years old
* Elementary education or above
* Able to communicate
* American Society of Anesthesiologists (ASA) physical status I-III
* Mini-mental State Examination (MMSE) scores ≥ 22 points

Exclusion Criteria:

* Preoperative delirium
* Severe mental diseases
* Autoimmune-illness, chronic infectious diseases, nervous system diseases and malignancies

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Eligible patients were scheduled to undergo elective orthopedics surgery under spinal anesthesia with an expected hospital stay of at least 3 days and received postoperative patient- controlled analgesia. Delirium was evaluated at the preoperative visit, then twice daily for 3 days following surgery. Cognition assessment was conducted at preoperative visit, 24 h after surgery and 72 h after surgery. Delirium assessments were performed before 10 AM and after 5 PM in the ward. The confusion assessment method (CAM) questionnaire and cognition assessment method for MMSE were performed by the qualified doctor who trained with CAM and MMSE training manual.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Confusion assessment method (CAM) score | Baseline (Before surgery)
  Positive CAM score means that the patient developed postoperative delirium. While negative CAM score means that the patient did not develop postoperative delirium.
CAM score | Postoperative day 1
  Positive CAM score means that the patient developed postoperative delirium. While negative CAM score means that the patient did not develop postoperative delirium.
CAM score | Postoperative day 2
  Positive CAM score means that the patient developed postoperative delirium. While negative CAM score means that the patient did not develop postoperative delirium.
CAM score | Postoperative day 3
  Positive CAM score means that the patient developed postoperative delirium. While negative CAM score means that the patient did not develop postoperative delirium.

SECONDARY OUTCOMES:
The level of systemic inflammation response index (SIRI) in peripheral blood. | Baseline (Before surgery)
  The SIRI was calculated as neutrophil count × monocyte count/lymphocyte count.
Mini-mental State Examination (MMSE) score | Baseline (Before surgery)
  MMSE score ranges from 0 to 30 and higher score means better outcome.
MMSE score | postoperative day 1
  MMSE score ranges from 0 to 30 and higher score means better outcome.
MMSE score | postoperative day 3
  MMSE score ranges from 0 to 30 and higher score means better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China